CLINICAL TRIAL: NCT02335580
Title: Effect of Portal Vein Thrombosis on the Prognosis of Liver Cirrhosis: A Single-center, Prospective, Cohort Study
Brief Title: Effect of Portal Vein Thrombosis on the Prognosis of Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Dr., General Hospital of Shenyang Military Region
Other Study IDs: PVT-LC Prognosis
Record Dates: First submitted 2015-01-07; First posted 2015-01-12 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Liver Cirrhosis; Portal Vein; Venous Thrombosis; Varicose Veins; Hemorrhage
Keywords: Prognosis
MeSH Terms: conditions — Liver Cirrhosis; Venous Thrombosis; Varicose Veins; Hemorrhage | interventions — Somatostatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Somatostatin and its analogs — Somatostatin and/or octreotide will be intravenously infused.
Procedure: Endoscopic sclerotherapy, endoscopic variceal ligation, endoscopic tissue glue injection — Endoscopic sclerotherapy, endoscopic variceal ligation, and/or endoscopic tissue glue injection will be performed based on the endoscopists' choice.

SUMMARY:
The prevalence of portal vein thrombosis (PVT) in patients with liver cirrhosis is 5-20%. Current evidence regarding the effect of portal vein thrombosis on the prognosis of cirrhotic patients remains under debate. Considering that PVT potentially elevates the portal pressure and thereby increase the risk of variceal bleeding, we focus on the patients with high-risk varices and variceal bleeding as the study population. Thus, the main goals are to analyze the effect of PVT on the incidence of first variceal bleeding in patients without any prior bleeding history but with high-risk varices, the incidence of recurrent variceal bleeding in patients with a history of variceal bleeding, and the treatment failure rate of variceal bleeding in patients with acute variceal bleeding. Certainly, the survival is also observed in all patients.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of liver cirrhosis.
2. Patients should be diagnosed with high-risk varices endoscopically, or a prior history of variceal bleeding, or an episode of acute variceal bleeding.
3. Patients agreed to undergo endoscopy to evaluate the presence and severity of varices.
4. Patients agreed to undergo contrast-enhanced CT scans to evaluate the portal vein patency. But if an abdominal contrast-enhanced CT scans was performed within 3 months after admission, it was not necessarily repeated.

Exclusion Criteria:

1. Non-cirrhotic patients.
2. Malignancy.
3. Contrast-enhanced CT scans were neither feasible nor available.
4. Severe cardiopulmonary diseases.
5. Severe infectious diseases.
6. Pregnant or breastfeeding.
7. Allergic to contrast agents.
8. Poor adherence.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population should be the patients with a diagnosis with liver cirrhosis who were admitted to the Department of Gastroenterology of General Hospital of Shenyang Military Area.
Sampling Method: Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | 6-24 months
First bleeding | 0-24 months
  As for the patients without any prior history of bleeding but with high-risk varices, the first bleeding was observed.
Recurrent bleeding | 0-24 months
  As for the patients with a prior history of bleeding, the recurrent bleeding was observed.
Treatment failure rate of acute variceal bleeding | 5 days
  As for the patients with acute variceal bleeding, the 5-day treatment failure of acute bleeding was observed.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, General Hospital of Shenyang Military Area, Shenyang, Liaoning, China

REFERENCES:
- [Background] Qi X, Han G, Fan D. Management of portal vein thrombosis in liver cirrhosis. Nat Rev Gastroenterol Hepatol. 2014 Jul;11(7):435-46. doi: 10.1038/nrgastro.2014.36. Epub 2014 Apr 1. PMID 24686266
- [Background] Qi X, Yang Z, Fan D. Spontaneous resolution of portal vein thrombosis in cirrhosis: where do we stand, and where will we go? Saudi J Gastroenterol. 2014 Sep-Oct;20(5):265-6. doi: 10.4103/1319-3767.141680. No abstract available. PMID 25253359
- [Background] Qi X, Wang J, Chen H, Han G, Fan D. Nonmalignant partial portal vein thrombosis in liver cirrhosis: to treat or not to treat? Radiology. 2013 Mar;266(3):994-5. doi: 10.1148/radiol.12122259. No abstract available. PMID 23431230
- [Background] Qi X, Han G, He C, Yin Z, Guo W, Niu J, Fan D. CT features of non-malignant portal vein thrombosis: a pictorial review. Clin Res Hepatol Gastroenterol. 2012 Dec;36(6):561-8. doi: 10.1016/j.clinre.2012.05.021. Epub 2012 Aug 9. PMID 22883835
- [Background] Qi X, Bai M, Yang Z, Yuan S, Zhang C, Han G, Fan D. Occlusive portal vein thrombosis as a new marker of decompensated cirrhosis. Med Hypotheses. 2011 Apr;76(4):522-6. doi: 10.1016/j.mehy.2010.12.007. Epub 2011 Jan 8. PMID 21216538
- [Background] Qi X, Han G, Wang J, Wu K, Fan D. Degree of portal vein thrombosis. Hepatology. 2010 Mar;51(3):1089-90. doi: 10.1002/hep.23397. No abstract available. PMID 19957371
- [Background] Qi X, Han G, Bai M, Fan D. Stage of portal vein thrombosis. J Hepatol. 2011 May;54(5):1080-2; author reply 1082-3. doi: 10.1016/j.jhep.2010.10.034. Epub 2010 Dec 5. No abstract available. PMID 21145872